CLINICAL TRIAL: NCT02328326
Title: Engaging Veterans and Family Supporters in PACT to Improve Diabetes Management
Brief Title: Caring Others Increasing EngageMent in PACT
Acronym: CO-IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 14-074
Record Dates: First submitted 2014-12-10; First posted 2014-12-31 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Diabetes
Keywords: Diabetes; diabetes self-management; patient activation; social support
MeSH Terms: conditions — Diabetes Mellitus; Patient Participation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CO-IMPACT (Experimental): patient and supporter (dyad) receive one coaching session on action planning, communicating with providers, navigation skills and support skills; preparation by phone before patients' primary care visits; after-visit summaries by mail; and biweekly automated phone calls to prompt action on new patient health concerns
  Interventions: Other: CO-IMPACT
- PACT (Active Comparator): patient and their health supporter (dyad) will receive PACT care for high-risk diabetes, which includes (at primary care team discretion): nurse care manager visits, diabetes education classes, chronic disease self-management groups, telehealth, clinical pharmacist visits
  Interventions: Other: PACT

INTERVENTIONS:
Other: CO-IMPACT — Primary care-integrated activation and social support intervention that provides tools and training in patient activation and effective support techniques for patients and their family supporter
  Arms: CO-IMPACT
Other: PACT — participants will receive PACT care for high-risk diabetes, which includes (at primary care team discretion): nurse care manager visits, diabetes education classes, chronic disease self-management groups, telehealth, clinical pharmacist visits
  Arms: PACT

SUMMARY:
This trial will compare two methods of increasing engagement in care and success in diabetes management, among patients with diabetes with high-risk features, who also have family members involved in their care.

DETAILED DESCRIPTION:
Background:

Veterans with diabetes must control cardiovascular risk factors in order to prevent disabling and life-threatening complications. However, despite system wide advances in diabetes quality of care, over 30% of VHA patients with diabetes continue to have uncontrolled blood pressure, hyperglycemia, or hyperlipidemia. The nationwide VA PACT (Patient-Aligned Care Teams) initiative seeks to provide patients comprehensive, team-based support for following diabetes care regimens. PACT's success, however, hinges on its ability to effectively engage patients in care. One relatively untapped resource for supporting engagement in PACT is patients' family and friends. Three out of four adults with diabetes reach out to an unpaid family member or friend (a 'Care Partner') for ongoing help with diabetes management. These supporters help patients with medication adherence, tracking home glucose measurements, maintaining a healthy eating plan, and often accompany patients to their medical visits. However, while PACT emphasizes the importance of family members as part of the care team, PACT does not have formal mechanisms to involve health supporters in PACT care. Health supporters report that, in order to be more effective, they need more information on patient's medical care plans, clear channels for communicating with PACT team members, and information on navigating PACT resources.

Objectives:

The overall objective of this randomized trial is to test a strategy to strengthen the capacity of supporters to help patients with high-risk diabetes engage in PACT care and successfully enact care plans.

The central hypothesis is that providing health care engagement tools to both Care Partners and patients will increase patient activation and improve management of diabetes complication risks.

Methods:

This is a randomized controlled trial evaluating an intervention (Caring Others Increasing EngageMent in PACT, or CO-IMPACT) designed to structure and facilitate health supporter involvement in PACT so that patients can become more actively engaged in PACT care. 240 patients with diabetes receiving PACT primary care who: 1) are at high risk for diabetes complications due to hyperglycemia OR high blood pressure and 2) have a health supporter involved in their care will be recruited along with their health supporter. Patient-supporter dyads are randomized to the CO-IMPACT intervention or usual PACT care for high-risk diabetes, for 12 months.

The intervention provides patient-supporter dyads: one coaching session on action planning, communicating with providers, navigation skills and support skills; preparation by phone before patients' primary care visits; after-visit summaries by mail; and biweekly automated phone calls to prompt action on new patient health concerns. CO-IMPACT builds on medical record-integrated patient activation tools in the PACT toolkit and is designed to be implementable within existing PACT nurse encounters.

Primary outcomes for this study include a validated measure of patient activation (Patient Activation Measure-13) and a cardiac event 5-year risk score designed for patients with diabetes (UKPDS Risk Engine). Secondary outcomes include patients' self-efficacy for diabetes self-care; diabetes self-management behaviors including medication adherence; diabetes distress; and glycemic and blood pressure control. Measures among supporters include supporter activation, use of effective support techniques, distress about patient's diabetes care, and caregiver burden. We are also measuring patient-supporter and patient-provider relationship quality, patient safety (e.g. hypoglycemia), utilization, potential moderators of intervention effect such as patient health literacy level, and facilitators and barriers to wider implementation.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria:

* Provide signed and dated informed consent form
* Plan to be be available for the duration of the study
* Male or female, age 30-70 years old
* Plan to get most diabetes care at recruiting VA primary care clinic over the subsequent 12 months
* Able to use telephone to respond to bi-weekly automated Interactive Voice Response (IVR) calls
* Be able to identify an adult family member or friend who is regularly involved in their health management or health care (involved with medications, managing sugars, coming to appointments, etc)
* Have a diagnosis of diabetes and be at high-risk for diabetes complications, defined as: (1) a diagnosis of diabetes based on encounter diagnoses from 1 inpatient or 2 outpatient encounters (OR a diabetes medication (at least one >3 month prescription from VA drug classes HS501 (insulin) or HS502, other than metformin), (2) have an assigned VAprimary care provider and at least 2 visits to VA primary care in the previous 12 months, (3) poor glycemic control (last HbA1C within 9 months >8%) OR poor blood pressure control (last BP 160/100 or mean 6 month BP >150/90)

Care Partner Inclusion Criteria:

* 21 years old or older
* Fluent in English
* Live in the United States

Exclusion Criteria:

Patient Exclusion Criteria:

* Expect to have >1 month gap in VA care in the 12 months following enrollment (e.g. snowbird travel).
* Plan to receive the majority of their care for diabetes mainly from a non-Primary Care provider in the 12 months following enrollment
* Have a VA resident/trainee as their main primary care provider
* Live in a nursing home OR assisted living
* Have significant cognitive impairment as measured by an Electronic Medical Record (EMR) diagnosis of Alzheimer's disease or dementia, or a score of <4 on the Callahan screener to identify cognitive impairment
* Need help with more than two basic activities of daily living (ADLs) as measured by the Katz Basic Activities of Daily Living Scale
* Do not speak English
* Have a life-limiting severe illness (such as stage renal disease [ESRD] requiring dialysis, chronic obstructive pulmonary disease (COPD) requiring oxygen, cancer undergoing active treatment, receiving palliative/hospice care)
* Are concurrently enrolled in another research study or clinical program, at time of enrollment, that could conflict with the current study's protocol (e.g. another diabetes management research intervention, or VA tele-buddy program involving frequent phone calls)
* Do not have a working phone or are not able to use a telephone to respond to automated IVR calls
* Currently Pregnant or planning to become pregnant at time of enrollment
* Have a serious mental illness or active substance abuse issue

Care Partner Exclusion Criteria:

* Receive pay for caring for the patient
* talks with patient about health less than two times per month
* Have significant cognitive impairment as measured by a score of 4 or less <4 on the Callahan screener to identify cognitive impairment
* Need help with more than two basic ADL as measured by the Katz Basic Activities of Daily Living Scale
* Have a life-limiting severe illness (such as end-stage renal disease requiring dialysis, chronic lung disease requiring oxygen, cancer undergoing active treatment, receiving palliative/hospice care)
* Ever told by a doctor they have dementia, schizophrenia, or manic depression

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2020-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie Rosland, MD MS, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Final dataset underlying publication resulting from this research will be shared upon request. Members of the scientific community can request a de-identified copy of the final dataset (i.e., dataset underlying any publication).
Access Criteria: Members of the scientific community should contact the PI. De-identified data may only be provided after requestors and data providers sign a standard federal agency Data Use Agreement.

REFERENCES:
- [Background] Rosland AM, Piette JD, Trivedi R, Kerr EA, Stoll S, Tremblay A, Heisler M. Engaging family supporters of adult patients with diabetes to improve clinical and patient-centered outcomes: study protocol for a randomized controlled trial. Trials. 2018 Jul 24;19(1):394. doi: 10.1186/s13063-018-2785-2. PMID 30041685
- [Result] Zupa MF, Lee A, Piette JD, Trivedi R, Youk A, Heisler M, Rosland AM. Impact of a Dyadic Intervention on Family Supporter Involvement in Helping Adults Manage Type 2 Diabetes. J Gen Intern Med. 2022 Mar;37(4):761-768. doi: 10.1007/s11606-021-06946-8. Epub 2021 Jul 8. PMID 34240285
- [Derived] Rosland AM, Piette JD, Trivedi R, Lee A, Stoll S, Youk AO, Obrosky DS, Deverts D, Kerr EA, Heisler M. Effectiveness of a Health Coaching Intervention for Patient-Family Dyads to Improve Outcomes Among Adults With Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2237960. doi: 10.1001/jamanetworkopen.2022.37960. PMID 36374502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 11/16/16 to 5/22/18. Eligible patient participants were identified from one of two participating VHA sites. Once identified, they received an introductory letter about the study and indicated interest by phone or mail.
Pre-assignment Details: None. All patient-supporter dyads who enrolled in the study were randomized to one of two study arms.
Groups:
- CO-IMPACT: patient and supporter (dyad) receive one coaching session on action planning, communicating with providers, navigation skills and support skills; preparation by phone before patients? primary care visits; after-visit summaries by mail; and biweekly automated phone calls to prompt action on new patient health concerns
  CO-IMPACT: Primary care-integrated activation and social support intervention that provides tools and training in patient activation and effective support techniques for patients and their family supporter
Period: Overall Study
Arm/Group | CO-IMPACT | PACT
Started | 246 (3 participant dyads withdrew before 6-month follow up. 3 more care partners withdrew and 1 died.) | 232 (1 participant dyad withdrew from the study between assignment to control arm and 6-month follow up.)
6-month Follow Up | 221 (We were unable to reach 15 participants. 1 patient died, 1 care partner withdrew before completion.) | 221 (We were unable to reach 9 participants. 1 patient died, 1 care partner withdrew before completion.)
Completed | 224 | 224
Not Completed | 22 | 8
Not completed — Withdrawal by Subject | 10 | 3
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CO-IMPACT | PACT | Total
Number analyzed (Participants) | 246 | 232 | 478
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Care Partner participant age was not collected in this study. Therefore median ages reflect only patient participants' median age.
  years
    Patient Participants: number analyzed (Participants) | 123 | 116 | 239
    Patient Participants | 62 [55 to 67] | 64 [52 to 68] | 64 [53 to 67]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants were recruited in patient-care partner dyads. As such, each row population has half as many participants analyzed as the total sample. For CO-IMPACT dyads, 246 total participants becomes 123 patient participants and 123 care partners. For PACT dyads, 232 becomes 116 and 116.
  Participants
    Patient Participants: number analyzed (Participants) | 123 | 116 | 239
    Patient Participants: Female | 6 | 2 | 8
    Patient Participants: Male | 117 | 114 | 231
    Care Partners: number analyzed (Participants) | 123 | 116 | 239
    Care Partners: Female | 14 | 10 | 24
    Care Partners: Male | 109 | 106 | 215
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants were recruited in patient-care partner dyads. As such, each row population has half as many participants analyzed as the total sample. For CO-IMPACT dyads, 246 total participants becomes 123 patient participants and 123 care partners. For PACT dyads, 232 becomes 116 and 116.
  Participants
    Patient Participants: number analyzed (Participants) | 123 | 116 | 239
    Patient Participants: Hispanic or Latino | 10 | 4 | 14
    Patient Participants: Not Hispanic or Latino | 112 | 112 | 224
    Patient Participants: Unknown or Not Reported | 1 | 0 | 1
    Care Partners: number analyzed (Participants) | 123 | 116 | 239
    Care Partners: Hispanic or Latino | 6 | 5 | 11
    Care Partners: Not Hispanic or Latino | 117 | 111 | 228
    Care Partners: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants were recruited in patient-care partner dyads. As such, each row population has half as many participants analyzed as the total sample. For CO-IMPACT dyads, 246 total participants becomes 123 patient participants and 123 care partners. For PACT dyads, 232 becomes 116 and 116.
  Participants
    Patient Participants: number analyzed (Participants) | 123 | 116 | 239
    Patient Participants: American Indian or Alaska Native | 6 | 0 | 6
    Patient Participants: Asian | 0 | 0 | 0
    Patient Participants: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Patient Participants: Black or African American | 12 | 18 | 30
    Patient Participants: White | 90 | 92 | 182
    Patient Participants: More than one race | 6 | 0 | 6
    Patient Participants: Unknown or Not Reported | 9 | 5 | 14
    Care Partners: number analyzed (Participants) | 123 | 116 | 239
    Care Partners: American Indian or Alaska Native | 1 | 0 | 1
    Care Partners: Asian | 0 | 1 | 1
    Care Partners: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Care Partners: Black or African American | 10 | 16 | 26
    Care Partners: White | 103 | 92 | 195
    Care Partners: More than one race | 5 | 2 | 7
    Care Partners: Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 246 | 232 | 478
Insulin Use among Patient Participants [Count of Participants; unit: Participants] — Population: Insulin Use was only collected for patient participants, but not their care partners.
  Participants
    number analyzed (Participants) | 123 | 116 | 239
    (all) | 78 | 64 | 142
PAM-13 Cutoff [Count of Participants; unit: Participants] — (Patient Activation Measure-13) - theoretical range of potential values (0,100), higher scores mean a better outcome, mean is computed for the difference in PAM scores from baseline to twelve months, among patient participants Population: Participants were recruited in patient-care partner dyads. As such, each row population has half as many participants analyzed as the total sample. For CO-IMPACT dyads, 246 total participants becomes 123 patient participants and 123 care partners. For PACT dyads, 232 becomes 116 and 116.
  Participants
    PAM-13 Prorated Score <40: number analyzed (Participants) | 123 | 116 | 239
    PAM-13 Prorated Score <40 | 55 | 65 | 120
    PAM-13 Prorated Score >40: number analyzed (Participants) | 123 | 116 | 239
    PAM-13 Prorated Score >40 | 68 | 51 | 119
Care Partner Lives with Patient Participant [Count of Participants; unit: Participants] — Population: This measure is specific to the care partners only.
  Participants
    number analyzed (Participants) | 123 | 116 | 239
    (all) | 86 | 82 | 168
Patient Baseline Patient Activation Measure (PAM-13) [Mean (Standard Deviation); unit: units on a scale] — (Patient Activation Measure-13) - theoretical range of potential values (0,100), higher scores mean a better outcome, mean score is computed at baseline among patient participants Population: This measure includes data from Patient Participants only
  units on a scale
    number analyzed (Participants) | 123 | 116 | 239
    (all) | 62.8 (11.2) | 59.8 (12.6) | 61.3 (12.0)
Baseline UKPDS 5-Year Cardiac Risk Score [Mean (Standard Deviation); unit: units on a scale] — United Kingdom Prospective Diabetes Study Risk Engine, among patient participants only, theoretical range is 0 to 100%, lower score equals a lower likelihood of an acute cardiac event over the next 5 years. Scores incorporate the individuals' level of HbA1c, blood pressure, cholesterol, and smoking status. Mean is computed at baseline among patient participants. Population: UKPDS Score only assessed among patient participants.
  units on a scale
    number analyzed (Participants) | 123 | 116 | 239
    (all) | 14.7 (10.0) | 13.6 (9.9) | 14.2 (9.9)
Enrolled at Hospital-based clinic (vs. community clinic site) [Count of Participants; unit: Participants] — Population: This measure is only among patient participants.
  Participants
    number analyzed (Participants) | 123 | 116 | 239
    (all) | 78 | 87 | 165

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Activation, as Measured by Patient Activation Measure - 13
Description: Patient Activation Measure-13. Range of potential values (0,100), higher scores mean a better outcome, Outcome is the participant's difference in the measure between baseline and 12 months, among patient participants
Time Frame: Baseline to 12 months
Population: This outcome was assessed only among patient participants and not among family supporters, so sample size for these analyses are approximately half of the total study population.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CO-IMPACT: patient and supporter (dyad) receive one 45-minute coaching session on understanding care partner's role; understanding patient's diabetes-related health information; patient engagement (action planning, communicating with providers); effective supporter techniques; and how to navigate VA resources (explain what PACT team is, how to reach them, VA diabetes-related programs). Throughout the year of the CO-IMPACT intervention, patient-supporter dyads receive preparation by phone before patients' primary care visits; after-visit summaries by mail; and biweekly automated phone calls to prompt action on new patient health concerns
  CO-IMPACT: Primary care-integrated activation and social support intervention that provides tools and training in patient activation and effective support techniques for patients and their family supporter.
- PACT: patient and their health supporter (dyad) will receive PACT care for high-risk diabetes, which follow VA/DoD diabetes management guidelines. At the primary care team's discretion, patients in PACT may also receive: nurse care manager visits, diabetes education classes, chronic disease self-management groups, telehealth, clinical pharmacist visits. Participants will also be given access to the CO-IMPACT educational information on general diabetes management in web or hardcopy format.
  PACT: participants will receive PACT care for high-risk diabetes, which may include (at primary care team discretion): nurse care manager visits, diabetes education classes, chronic disease self-management groups, telehealth, and clinical pharmacist visits.
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 123 | 116
units on a scale | 2.94 (9.86) | 1.78 (10.84)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in PAM is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' PAM score compared to patient participants in PACT; Test type: Superiority; p = 0.048, Regression, Linear; Model was adjusted for baseline value of PAM, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 2.60, 95% CI 2-sided [0.02 to 5.18] — Net difference defined as 12 months minus baseline

2. Primary Outcome: Change in Cardiac Event 5-year Risk Score, as Measured by UKPDS Risk Engine
Description: UKPDS Risk Engine, among patient participants only, range is 0 to 100% risk of cardiac event over the next 5 years. Lower score equals a better outcome. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 123 | 116
units on a scale | 0.14 (6.77) | -0.73 (6.51)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in ukpds 5 year risk score is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly decrease patient participants' 5-year cardiovascular event risk; Test type: Superiority; p = 0.32, Regression, Linear; Model adjusted for baseline value of ukpds, insulin use, site, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.9, 95% CI 2-sided [-0.87 to 2.67] — Net difference defined as 12 months minus baseline. Reference for comparison is PACT

3. Secondary Outcome: Change in Diabetes Self-Management Behavior - Healthy Eating
Description: Summary of Diabetes Self-Care Activities (SDSCA) - range of potential values for healthy eating subscale (0 - 7 days per week), higher scores mean better outcomes, among patient participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: The outcomes was assessed only among patient participants and not among family supporters, so sample size for these analyses are approximately half of the total study population. Only participants with complete baseline and 12 month data for the outcome were included in that outcome's analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 116 | 113
score on a scale | 1.12 (2.30) | 0.50 (2.54)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in Healthy Eating is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly change patient participants' Healthy Eating scores compared to patient participants in PACT; Test type: Superiority; p = 0.01, Regression, Linear; Model adjusted for BL value of Healthy Eating, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.71, 95% CI 2-sided [0.20 to 1.22] — Net difference defined as 12 months minus baseline

4. Secondary Outcome: Change in Glycemic Control
Description: Hemoglobin A1c, among patient participants. Common range is 4% to 14%, lower values indicate better outcomes. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of glycosylated hemoglobin
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 114 | 113
percent of glycosylated hemoglobin | -0.05 (1.38) | -0.28 (1.43)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in A1c is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly decrease patient participants' A1c score compared to patient participants in PACT; Test type: Superiority; p = 0.33, Regression, Linear; Model was adjusted for baseline value of A1c, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.17 to 0.51] — Net difference defined as 12 months minus baseline

5. Secondary Outcome: Change in Systolic Blood Pressure
Description: mmHg, Average of two readings done at each time point. Common physiologic range is 80mmHg - 220mmHg. Lower values indicate better outcomes, among patient participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 110 | 110
mmHg | -6.41 (1.75) | -2.46 (1.77)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in SBP is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly decrease patient participants' SBP score compared to patient participants in PACT; Test type: Superiority; p = 0.18, Regression, Linear; Model was adjusted for baseline value of SBP, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = -2.82, 95% CI 2-sided [-7.00 to 1.35] — Net difference defined as 12 months minus baseline

6. Secondary Outcome: Change in Diabetes Distress
Description: Problem Areas in Diabetes Scale (PAID) - range of potential values (0,20), higher scores indicate worse outcomes (greater diabetes-related emotional distress), among patient participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 114 | 111
score on a scale | -0.25 (4.06) | -0.62 (4.60)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in PAID is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' PAID score compared to patient participants in PACT; Test type: Superiority; p = 0.83, Regression, Linear; Model was adjusted for baseline value of PAID, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.95 to 1.19] — Net difference defined as 12 months minus baseline

7. Secondary Outcome: Change in Activation in Health Encounters
Description: Perceived Efficacy in Patient-Physician Interactions (PEPPI-5) - range of potential values (5, 25), higher scores indicate better outcomes (higher perceived self-efficacy in patient-physician interactions), among patient participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 115 | 113
score on a scale | 0.23 (3.41) | 0.33 (4.01)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in PEPPI is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' PEPPI score compared to patient participants in PACT; Test type: Superiority; p = 0.79, Regression, Linear; Model was adjusted for baseline value of PEPPI, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.71 to 0.93] — Net difference defined as 12 months minus baseline

8. Secondary Outcome: Change in Non-Fasting Lipid Levels
Description: Total cholesterol mg/DL to HDL mg/DL Ratio, common range is 1-10, lower values indicate better outcomes, among patient participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 114 | 113
mg/dL | -0.11 (0.99) | -0.21 (1.01)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in Chol to HDL Ratio is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly decrease patient participants' Chol to HDL Ratio score compared to patient participants in PACT; Test type: Superiority; p = 0.21, Regression, Linear; Model adjusted for BL value of Cho to HDL Ratio, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Median Difference (Net) = 0.15, 95% CI 2-sided [-0.09 to 0.40] — Net difference defined as 12 months minus baseline

9. Secondary Outcome: Change in Patient Satisfaction With Healthcare System Support for Family Supporter
Description: Measured as percent of patient participants answering they were 'very satisfied' or 'satisfied' with healthcare system support for their Care Partner (family supporter)'s participation in their healthcare. Response options were 'very unsatisfied', 'unsatisfied', 'neither', 'satisfied', or 'very satisfied'. Increase in proportion of 'very satisfied' or 'satisfied' indicates better outcomes (higher satisfaction), among patient participants.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 115 | 111
Participants
  Number moving from not satisfied/neither to satisfied | 35 | 20
  Those not changing or getting worse | 80 | 91

10. Secondary Outcome: Change in Supporter Use of Autonomy-Supportive Communication
Description: Important Other Climate Questionnaire (IOCQ) - patient rating of supporter communication. Range of potential values (1,7), higher scores indicate better outcomes (higher patient perception of supporter use of autonomy supportive communication), among patient participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 110 | 113
score on a scale | 0.27 (0.93) | 0.05 (0.94)
Statistical Analysis 1: Comparison: CO-IMPACT; The null hypothesis was that change (baseline to 12 months) in IOCQ is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' IOCQ score compared to patient participants in PACT; Test type: Superiority; p = 0.01, Regression, Linear; Model was adjusted for baseline value of IOCQ, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.30, 95% CI 2-sided [0.08 to 0.53] — Net difference defined as 12 months minus baseline

11. Secondary Outcome: Change in Smoking Status
Description: Global Adult Tobacco Survey, values include 'current smoker', 'former smoker', or 'never smoker'. Change from current to former smoker over 12 months indicates a better outcome. Measured among patient participants.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 115 | 113
Participants
  Changed from active smoker at baseline to non-smoker at 12 months | 2 | 3
  Changed from non-smoker at baseline to smoker at 12 months | 1 | 5
  No change | 112 | 105
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; Test type: Equivalence — Equivalent distribution among categories; p = 0.17, Chi-squared; difference in count = -1; Difference in count of those who stopped smoking in CO-IMPACT vs. those who stopped smoking in PACT

12. Secondary Outcome: Change in Diabetes Self-Management Behavior - Physical Activity
Description: Summary of Diabetes Self-Care Activities (SDSCA) - range of potential values for physical activity subscale (0-7 days per week), higher scores mean better outcome, among patient participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 115 | 113
score on a scale | 0.09 (2.46) | 0.46 (2.13)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in Physical activity is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' Physical activity score compared to patient participants in PACT; Test type: Superiority; p = 0.87, Regression, Linear; Model adjusted for BL value of Physical Activity, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.56 to 0.47] — Net difference defined as 12 months minus baseline

13. Secondary Outcome: Change in Diabetes Self-Management Behavior - Blood Sugar Home Testing
Description: Summary of Diabetes Self-Care Activities (SDSCA) - range of potential values (0-7 days per week), higher scores mean better outcome, among patient participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: The outcome was assessed only among patient participants and not among family supporters, so sample size for these analyses are approximately half of the total study population. Only participants with complete baseline and 12 month data for the outcome were included in that outcome's analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 101 | 94
score on a scale | 0.17 (1.75) | 0.19 (1.80)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in Blood Sugar Home Testing is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' Blood Sugar Home Testing score compared to patient participants in PACT; Test type: Superiority; p = 0.31, Regression, Linear; Model adjusted for BL value of Blood Sugar Home Testing, insulin use, randomization strat. variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.22 to 0.68] — Net difference defined as 12 months minus baseline

14. Secondary Outcome: Change in Diabetes Self-Management Behavior - Blood Pressure Home Testing
Description: as for outcome 13
Time Frame: Baseline to 12 months
Population: This outcome was assessed only among patient participants and not among family supporters, so sample size for these analyses are approximately half of the total study population. The outcomes was assessed only among patient participants and not among family supporters, so sample size for these analyses are approximately half of the total study population. Only participants with complete baseline and 12 month data for the outcome were included in that outcome's analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 75 | 62
score on a scale | 0.51 (2.52) | 0.48 (1.88)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in Blood Pressure Home Testing is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' Blood Pressure Home Testing score compared to patient participants in PACT; Test type: Superiority; p = 0.87, Regression, Linear; Model adjusted for BL value of Blood Pressure Home Testing, insulin use, randomization strat. variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.76 to 0.89] — Net difference defined as 12 months minus baseline

15. Secondary Outcome: Change in Diabetes Self-Management Behavior - Take Oral Meds as Prescribed
Description: as for outcome 13
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 99 | 96
score on a scale | 0.14 (1.17) | 0.23 (1.30)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in Take Oral Meds as Prescribed is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' Take Oral Meds as Prescribed score compared to patient participants in PACT; Test type: Superiority; p = 0.56, Regression, Linear; Model adjusted for BL value of Take Oral Meds as Prescribed, insulin use, randomization strat variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.42 to 0.23] — Net difference defined as 12 months minus baseline

16. Secondary Outcome: Change in Diabetes Self-Management Behavior - Take Insulin as Prescribed
Description: as for outcome 13
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 73 | 61
score on a scale | 0.14 (1.34) | 0.48 (2.08)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in Take Insulin as prescribed is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' Take Insulin as Prescribed compared to patient participants in PACT; Test type: Superiority; p = 0.67, Regression, Linear; Model adjusted for baseline value of Take Insulin as Prescribed, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.26 to 0.41] — Net difference defined as 12 months minus baseline

17. Secondary Outcome: Change in Diabetes Self-Management Behavior - Check Feet
Description: as for outcome 13
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 115 | 113
score on a scale | 0.72 (2.06) | 0.72 (2.26)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; Test type: Superiority — The null hypothesis was that change (baseline to 12 months) in Foot Care is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' Foot Care score compared to patient participants in PACT; p = 0.29, Regression, Linear; Model was adjusted for baseline value of Foot Care, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Median Difference (Net) = 0.26, 95% CI 2-sided [-0.22 to 0.75]; Net difference defined as 12 months minus baseline

18. Other Pre Specified Outcome: Change in Diabetes Self-Efficacy
Description: Adapted Stanford Chronic Disease self-efficacy scale, among patient participants. Range of potential values (1,10), higher score indicates higher self-efficacy. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 115 | 113
score on a scale | 0.26 (1.38) | 0.23 (1.48)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in SE is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly change patient participants' SE scores compared to patient participants in PACT; Test type: Superiority; p = 0.01, Regression, Linear; Model was adjusted for baseline value of SE, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.40, 95% CI 2-sided [0.09 to 0.71] — Net difference defined as 12 months minus baseline

19. Other Pre Specified Outcome: Change in Supporter Self-Efficacy for Helping With Diabetes Care
Description: Adapted Stanford Chronic Disease self-efficacy scale, among family supporter participants. Range of potential values (1,10), higher score indicates higher self-efficacy. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 108 | 110
score on a scale | 0.19 (1.77) | 0.29 (1.83)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in Lorig_CP is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' Lorig_CP score compared to patient participants in PACT; Test type: Superiority; p = 0.67, Regression, Linear; Model was adjusted for baseline value of Lorig_CP, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.34 to 0.55] — Net difference defined as 12 months minus baseline

20. Other Pre Specified Outcome: Change in Caregiver Burden
Description: Caregiver Strain Index - range of potential values (0,13), higher scores (7 or more) mean worse outcomes, among family supporter participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 108 | 108
score on a scale | 0.18 (3.77) | -0.54 (3.30)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in CSIS is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' CSIS score compared to patient participants in PACT; Test type: Superiority; p = 0.53, Regression, Linear; Mean Difference (Net) = 0.28, 95% CI 2-sided [-0.60 to 1.16] — Net difference defined as 12 months minus baseline

21. Other Pre Specified Outcome: Change in Supporter Distress About Patient Participant's Diabetes
Description: Adapted Problem Areas In Diabetes Scale (PAID) - range of potential values (0,20), higher scores indicate worse outcomes (greater diabetes-related emotional distress), among family supporter participants. Outcome is the participant's difference in the measure between baseline and 12 months.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO-IMPACT | PACT
Number analyzed (Participants) | 107 | 108
score on a scale | -0.50 (3.57) | -1.08 (3.71)
Statistical Analysis 1: Comparison: CO-IMPACT vs PACT; The null hypothesis was that change (baseline to 12 months) in PAID_CP is the same for CO-IMPACT (intervention) compared to PACT (control). The alternative hypothesis is that that COIMPACT will significantly increase patient participants' PAID_CP score compared to patient participants in PACT; Test type: Superiority; p = 0.50, Regression, Linear; Model was adjusted for baseline value of PAID_CP, insulin use, randomization stratification variables: care partner not in home and PAM cutoff of 40; Mean Difference (Net) = 0.32, 95% CI 2-sided [-0.61 to 1.25] — Net difference defined as 12 months minus baselineNet difference defined as 12 months minus baseline

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the year participants were enrolled in the study. All participants participated between the dates of 01/03/17 to 06/03/19.
Description: Definitions of adverse event and serious adverse event used by study team were consistent with the clinicaltrials.gov definitions. Adverse events were collected when self-reported by participants or family members when study staff reached out to schedule or conduct intervention components or assessment visits.
Arm/Group | CO-IMPACT | PACT
All-Cause Mortality (participants affected / at risk) | 2/246 | 1/232
Serious Adverse Events (participants affected / at risk) | 29/246 | 2/232
Other Adverse Events (participants affected / at risk) | 0/246 | 0/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CO-IMPACT (N=246) | PACT (N=232)
Cardiac Events (Cardiac disorders) | 6 (6) | 0 (0) — 3 patient participants (PT) had heart attacks; 1 PT in hospital for "heart issues"; 1 PT hospitalized CHF; 1 PT hospitalized arrythmia
Vascular Issues (Vascular disorders) | 3 (3) | 1 (1) — 2 patient participants (PT) hospitalized for high blood pressure (1 intervention, 1 control); 1 PT hospitalized low blood pressure; 1 PT in emergency room for blood clot
Infection (Infections and infestations) | 4 (4) | 0 (0) — 1 patient participant (PT) hospitalized due to infection; 1 PT hospitalized for sepsis; 1 PT eye infection; 1 PT sinus infection.
Surgeries (Surgical and medical procedures) | 4 (4) | 0 (0) — 2 patient participants (PT) had lower limb amputations; 1 PT hand injury & surgery; 1 PT emergency intestinal surgery
Injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) — 1 patient participant (PT) broken bone in lower limb; 1 PT car accident; 2 PTs broken bones or dislocations upper limbs
Stroke (Nervous system disorders) | 4 (4) | 0 (0) — 4 patient participants (PT) had strokes, all withdrew. 2 PT hospitalized for passing out, one had renal failure also; 1 PT in and out of hospital since stroke; 1 PT withdrawn by Care partner because not cognitively present
General Diagnoses, Hospitalizations (General disorders) | 2 (2) | 1 (1) — 1 Control patient participant (PT) admitted to hospital (no reason provided ; 1 PT diagnosed cancer
Social Circumstances (Social circumstances) | 1 (1) | 0 (0) — 1 PT lost housing
Multiple Issues (General disorders) | 1 (1) | 0 (0) — One Patient participant had a stroke, kidney stones

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT02328326/Prot_SAP_000.pdf